CLINICAL TRIAL: NCT07263854
Title: Effects of Lower Extremity Neuromuscular Facilitation on Gait, Balance and Fatigue in Patients With Multiple Sclerosis: A Randomized Controlled Study
Brief Title: Effects of Lower Extremity Neuromuscular Facilitation and Patients With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanko University (Other)
Responsible Party: Principal Investigator, Hakan Polat, dırector, Sanko University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: hakanpolat7
Record Dates: First submitted 2025-11-17; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Gait Balance; Balance; Fatigue Syndrome, Chronic
Keywords: multipl skleroz; balance; gait; fatigue
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Fatigue | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- working group (Experimental): Proprioceptive neuromuscular facilitation (PNF) exercises
  Interventions: Other: exercises
- control group (Experimental): strengthening exercises
  Interventions: Other: exercises

INTERVENTIONS:
Other: exercises — Each of the two groups was given exercise three days a week for six weeks.

SUMMARY:
Objective: This study aimed to investigate the effects of lower extremity Proprioceptive Neuromuscular Facilitation (PNF) exercises on balance, gait, and fatigue in patients with Multiple Sclerosis (MS).

Method: Twenty-six MS patients (18 women, 8 men) were included in the study. Participants were divided into two groups. The study group (n=13) underwent lower extremity Proprioceptive Neuromuscular Facilitation exercises, while the control group (n=13) underwent lower extremity strengthening exercise training three days a week for six weeks. Static balance, tandem stance test, dynamic balance, walking with the 4-step square test, walking with the 25-step test, and fatigue were assessed twice, before and after treatment, using the fatigue severity scale.

DETAILED DESCRIPTION:
This study was conducted as a randomised, parallel-group, single-blind clinical trial in accordance with the CONSORT (Consolidated Standards of Reporting Trials) Guidelines. Ethical approval was obtained from the SANKO University Non-Interventional Clinical Research Ethics Committee (2024/11-5).

MS patients who volunteered from the SANKO University Faculty of Medicine Neurology Clinic were included in the study. Inclusion criteria were (i) diagnosis of Relapsing-Remitting Multiple Sclerosis (RRMS) according to the 2017 McDonald criteria, (ii) age 18-65, (iii) Expanded Disability Status Scale (EDSS) score of 4 or below, (iv) no relapse in the last 6 months. Exclusion criteria were (i) a history of lower extremity trauma within the last year, (ii) a history of known chronic neurological disorders, (iii) any contraindication to exercise, and (iv) cognitive impairment as defined by a mini-mental test (score below 24).

The required sample size for the study was determined using a power analysis performed with the G-Power 3.1* programme. The analysis resulted in a medium effect size for between-group comparisons at a 5% significance level (Type I error probability, α=0.05) and 85% statistical power (1-β=0.85), at least 11 participants were needed in each group to detect a medium effect size (Cohen's d ≈ 0.5) in between-group comparisons. A total of 26 participants, 13 in each of the Experimental and Control groups, were included in the study, and this number met the minimum sample size determined by the power analysis.

Forty patients diagnosed with MS were invited to participate in the study, but those who voluntarily withdrew or never started the study (n = 14) were excluded. The study was completed with 26 patients: 13 in the Study group (nine women, four men) and 13 in the Control group (nine women, four men). A minimisation method was used to balance the gender and clinical course of the participants, and a total of 26 patients were randomly assigned to the Study Group (PNFG, n:13) and the Control Group (CG, n:13) . The researcher responsible for randomisation did not participate in data collection or data analysis.

All patients' demographic information (age, gender, body mass index) and disease characteristics (disease duration and EDSS) were recorded. Subsequently, participants' walking, balance, and fatigue status were assessed. Assessments and treatment were conducted at the same time and in the same environment but on different days. Assessments were conducted with rest periods to eliminate fatigue and other potential issues. Two researchers, blinded to randomisation, assessed all patients twice: at baseline (BL) and six weeks later (WL). The physiotherapists administering the treatments did not participate in the assessments. Assignment was concealed from patients until after the baseline assessment. Patients were asked not to discuss their interventions with the assessors during the final assessment. Walking was assessed using a 25-step walking test, balance was assessed statically using a tandem stance test and dynamically using a four-step square test, and fatigue was assessed using a fatigue severity scale.

ELIGIBILITY:
Inclusion Criteria:

* (i) Having been diagnosed with Relapsing-Remitting Multiple Sclerosis (RRMS) according to the 2017 McDonald criteria (Thompson, Banwell et al. 2018), (ii) Aged 18-65 years, (iii) Expanded Disability Status Scale (EDSS) score of 4 or below, (iv) No relapses in the past 6 months.

Exclusion Criteria:

* (i) Having a history of trauma to the lower extremities within the last year, (ii) having a known history of other chronic neurological disorders, (iii) having any contraindications to exercise, (iv) cognitive impairment as defined by a mini-mental test (scoring below 24 points).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-09-16 (Actual)

PRIMARY OUTCOMES:
static balance | 6 weeks
  tandem stance test
dynamic balance | 6 weeks
  four-square test
gait | 6 weeks
  25-step walking test
fatigue | 6 weeks
  Fatigue Severity Scale (fSS): The **Fatigue Severity Scale (FSS)** is a 9-item measure that assesses the severity of fatigue, with each item scored on a scale of 1-7. The average score on the scale is typically considered. **A low FSS score (1.0-3.9)** indicates mild fatigue that does not significantly affect daily life; the individual generally has normal energy levels, and fatigue does not restrict work or social life. A **high FSS score (4.0-7.0)** indicates that fatigue is markedly excessive and negatively affects daily activities; it is consistent with decreased energy, difficulty performing activities, and fatigue seen in chronic illnesses. Clinically, an average score of **4 or above** is considered **significant fatigue**, while a score below 4 is considered **low fatigue**.

CONTACTS AND LOCATIONS:
Locations (1):
- Sanko Unıversıty, Gaziantep, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No